CLINICAL TRIAL: NCT02751983
Title: ACT for Life: a Brief Intervention for Maximizing Recovery After Suicidal Crises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2048-P; I21RX002048-01 (NIH)
Record Dates: First submitted 2016-04-21; First posted 2016-04-26 (Estimated); Results first posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Suicide; Psychiatric Rehabilitation
Keywords: Suicide; Psychiatric Rehabilitation; Acceptance and Commitment Therapy; Brief Psychotherapy; Inpatients
MeSH Terms: conditions — Suicide | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment as usual plus ACT (Experimental): Participants in this condition will be enrolled in the ACT for Life intervention and still able to engage in treatment as usual.
  Interventions: Behavioral: ACT for Life; Other: Treatment as usual
- Treatment as usual (Active Comparator): Participants in this condition will not be enrolled in ACT for Life, but will continue to participate in treatment as usual (e.g., inpatient and outpatient mental health care).
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: ACT for Life — A novel protocol detailing the application of Acceptance and Commitment Therapy (ACT) to recovery from suicidal crises. Consists of three modules designed to be delivered in three to four 60-minute individual talk therapy sessions. Nearly all of the metaphors and experiential exercises are adaptations of core ACT techniques included in various empirically-supported applications of ACT to other health conditions. Additionally, the adjunctive intervention is designed to augment safety planning (a hierarchical list of strategies to recognize and cope with a suicidal crisis).
  Arms: Treatment as usual plus ACT
Other: Treatment as usual — All participants will be able to engage in treatment as usual. Psychiatric inpatient care typically consists of behavioral mental health group and/or individual therapy and pharmacological treatment. Outpatient care is offered upon discharge. This typically consists of both group and individual therapy and medication management.

SUMMARY:
An estimated 20 Veterans kill themselves every day. Suicide prevention literature and public health policy both call for treatment targeting high-risk populations, such as Veterans hospitalized due to suicidal intent and/or attempts. Psychiatric hospitalization is a critical opportunity to provide treatment to reduce the risk of suicide and lay the groundwork for functional recovery. Yet, there are no interventions specifically for suicide prevention that meet Veterans Health Affairs' quality recommendations requiring the provision of evidence-based, recovery-oriented psychotherapy, which are also feasible to use during a typical inpatient stay. The proposed study seeks to take a first step toward filling this gap. In consultation with experts in the field, the authors have developed a protocol applying a recovery-oriented, evidence-based treatment approach to Veteran inpatient care. The proposed pilot study will provide critical information to inform final revisions of the treatment manual and research design for a future study evaluating the efficacy of the intervention.

DETAILED DESCRIPTION:
Psychiatric hospitalization presents a critical opportunity for delivering targeted treatment to reduce suicide risk and promote functional recovery. Yet, there are no suicide-specific empirically-supported interventions that can be feasibly delivered during a typical Veterans Health Affairs (VHA) inpatient stay. Although VHA now requires the provision of evidence-based, recovery-oriented inpatient psychotherapy, extant empirically-supported interventions for patients at high risk of suicide were developed for use in outpatient settings and are too time- and resource-intensive to implement as intended in inpatient psychiatric settings, where shorter lengths of stay are expected. Furthermore, these interventions focus nearly entirely on preventing suicidal behavior without also targeting functional recovery. Similarly, inpatient psychiatric treatment has traditionally focused on medical management of acute illness, not on improving patient functioning. Preventing suicide during a crisis is only a short-term solution if the investigators fail to assist patients in understanding how they can rebuild a life they deem worth living. Given that approximately 50% of inpatients do not engage in recommended outpatient mental health care and are at the highest risk of death by suicide, it is vital that inpatient care promote functional recovery. The ideal brief intervention for Veterans at risk for suicide needs to reduce risk of suicidal behavior while simultaneously fostering recovery.

Acceptance and Commitment Therapy (ACT) is a recovery-oriented, psychosocial treatment approach ideally suited for utilization among Veterans hospitalized for suicide risk. ACT teaches psychological skills to handle painful thoughts, emotions, and sensations, but rather than focusing on symptom reduction, ACT directly targets functional recovery by assisting patients in identifying and engaging in value-consistent behaviors despite the potential for distress. There are no brief, ACT-based, transdiagnostic treatment protocols designed to address suicide risk. In order to fill this gap, the investigators consulted with leading experts in ACT to develop and manualize "ACT for Life", a brief, transdiagnostic, recovery-oriented intervention for Veterans hospitalized due to suicide risk. The ACT for Life manual details the application of ACT to recovery from suicidal crises and consists of three modules, [designed to be utilized in three to four 60-minute individual sessions.] This two arm, randomized, controlled pilot study will provide critical information to inform final revisions to the treatment manual and research design for a future efficacy study of ACT for Life. Veterans who enroll in the study will be randomized to: (a) treatment as usual or (b) treatment as usual plus ACT. The specific aims of this study are to: (1) Determine the acceptability of ACT for Life. (2) Determine the feasibility of the study design and research procedures. (3) Characterize participants' psychosocial functioning and self-directed violence using candidate outcome measures for a future efficacy trial. All participants will complete a baseline assessment, and follow-up assessments one and three months after hospital discharge. Participants in the ACT group will also complete a post-treatment assessment on acceptability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for Veterans Health Administration care
* Age 18-89
* Currently hospitalized due to suicide risk
* Willing to be randomized and participate in the two conditions

Exclusion Criteria:

* Inability to provide informed consent
* Inability to complete study measures, e.g.:

  * due to significant acute intoxication/withdrawal symptoms
  * mania
  * psychosis
  * aggression
  * catatonia
  * cognitive impairment
* membership in vulnerable population, e.g.:

  * prisoners

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Michael Barnes, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6 participants (1 Treatment as Usual (TAU), 5 TAU plus ACT (ACT)), were enrolled in a "pilot to the pilot" phase of the current study. Clinicians were trained based on the first 5 ACT participants and qualitative feedback was used to revise the ACT for Life manual prior to enrolling an additional 70 participants who were randomized to ACT or TAU.
Groups:
- Treatment as Usual Plus ACT: Participants in this condition will be enrolled in the ACT for Life intervention and still able to engage in treatment as usual.
  ACT for Life: A novel protocol detailing the application of Acceptance and Commitment Therapy (ACT) to recovery from suicidal crises. Consists of three modules designed to be delivered in three to four 60-minute individual talk therapy sessions. Nearly all of the metaphors and experiential exercises are adaptations of core ACT techniques included in various empirically-supported applications of ACT to other health conditions. Additionally, the adjunctive intervention is designed to augment safety planning (a hierarchical list of strategies to recognize and cope with a suicidal crisis).
  Treatment as usual: All participants will be able to engage in treatment as usual. Psychiatric inpatient care typically consists of behavioral mental health group and/or individual therapy and pharmacological treatment. Outpatient care is offered upon discharge.
Period: Baseline and Randomization
Arm/Group | Treatment as Usual Plus ACT | Treatment as Usual
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0
Period: Treatment
Arm/Group | Treatment as Usual Plus ACT | Treatment as Usual
Started | 35 | 35
Completed | 31 | 35
Not Completed | 4 | 0
Not completed — Stopped ACT, but Remained in study | 2 | 0
Not completed — Discharged prior to beginning ACT | 2 | 0
Period: Post-Treatment Assessment
Arm/Group | Treatment as Usual Plus ACT | Treatment as Usual
Started | 35 | 0
Completed | 30 | 0
Not Completed | 5 | 0
Not completed — Lost to Follow-up | 5 | 0
Period: One-Month Follow-Up Assessments
Arm/Group | Treatment as Usual Plus ACT | Treatment as Usual
Started | 35 | 35
Completed | 21 | 23
Not Completed | 14 | 12
Not completed — Lost to Follow-up | 14 | 12
Period: Three-Month Follow-Up Assessments
Arm/Group | Treatment as Usual Plus ACT | Treatment as Usual
Started | 35 | 35
Completed | 23 | 19
Not Completed | 12 | 16
Not completed — Lost to Follow-up | 12 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual Plus ACT | Treatment as Usual | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 31 | 65
  >=65 years | 1 | 4 | 5
Age, Continuous [Median (Full Range); unit: years] | 42 [22 to 70] | 49 [27 to 73] | 47 [22 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 30 | 27 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 22 | 21 | 43
  Race: Black | 3 | 4 | 7
  Race: Native American/Alaskan native | 0 | 2 | 2
  Race: Asian | 1 | 1 | 2
  Race: Pacific Islander | 1 | 0 | 1
  Race: Multiracial | 5 | 6 | 11
  Race: Other | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 35 | 70
Sexual Orientation [Count of Participants; unit: Participants]
  Gay/Lesbian/Queer | 1 | 3 | 4
  Bisexual | 1 | 0 | 1
  Heterosexual | 32 | 30 | 62
  Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Client Satisfaction Questionnaire - 8
Description: Self-report measure that will be used to assess participants' satisfaction with ACT for Life. Scale scores range from 8 to 32 with higher scores indicating greater satisfaction. For the purposes of the current study scores greater than or equal to 24 were considered acceptable. The number of participants scoring ≥ 24 is reported below.
Time Frame: Post-treatment (0-7 days after treatment completion)
Population: Post-treatment data were collected from participants who engaged in at least one ACT for Life session. 2 of the 35 ACT participants discharged from the hospital prior to receiving any treatment. 3 participants discharged prior to post-treatment assessment and were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual Plus ACT
Number analyzed (Participants) | 30
Participants | 28

2. Primary Outcome: Narrative Evaluation of Intervention Interview
Description: Semi-structured interview assessing each participants' perspective of the impact of the intervention, helpful and unhelpful components, and comparison to other interventions. Will be used to assess acceptability and inform revisions to the treatment manual. Qualitative Thematic Analysis was conducted. There are no objective data to report from this interview. Please contact the PI for reference to a manuscript with the qualitative results.
Time Frame: Post-treatment (0-7 days after treatment completion)
Population: as for outcome 1
Measure: Number; unit: participants analyzed
Arm/Group | Treatment as Usual Plus ACT
Number analyzed (Participants) | 30
participants analyzed | 30

3. Primary Outcome: Reasons for Termination (Client and Therapist Versions)
Description: Self-report scale which assesses the impact of 19 common reasons why patients terminate therapy. Will be used to assess treatment acceptability. These participants reported reasons for termination of ACT, but this did not produce quantitative data.
Time Frame: Post-treatment (0-7 days after treatment termination)
Population: Data reflects those who terminated the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual Plus ACT
Number analyzed (Participants) | 30
Participants | 2

4. Secondary Outcome: Outcome Questionnaire 45.2 (OQ-45)
Description: The Outcome Questionnaire 45.2 is a 45-item self-report scale that assesses symptom distress, interpersonal relationships, and social role (functioning in the workplace, school, and home) for the past week. The OQ-45 total score ranges from 0-180 with higher scores indicating greater distress and impairment. Scores of 63 or more generally indicate symptoms of clinical significance and changes of 14 points or more are typically considered a "reliable change."
Time Frame: Pre-treatment, One-Month Follow-Up, Three-Month Follow-Up
Population: The number of participants analyzed in row two and three differ from row one because the results are from different time points and some participants were lost to follow up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment as Usual Plus ACT | Treatment as Usual
Number analyzed (Participants) | 35 | 35
score on a scale
  Pre-treatment | 95.20 [85.87 to 104.53] | 105.14 [97.81 to 112.48]
  One-month Follow-up: number analyzed (Participants) | 20 | 22
  One-month Follow-up | 68.10 [56.68 to 79.52] | 88.55 [77.80 to 99.29]
  Three-month Follow-up: number analyzed (Participants) | 20 | 19
  Three-month Follow-up | 72.05 [57.90 to 86.20] | 89.11 [79.05 to 99.16]

5. Secondary Outcome: Valued Living Questionnaire (Used to Assess Change)
Description: Self-report measure that assesses participants' life values as well as the perceived consistency with which they have been living according to their values. Will be examined as a candidate outcome measure for a future efficacy trial. The reported "composite score" accounts for both importance and consistency (mean of the products of importance and consistency scores within each domain) to quantify the extent to which one is contacting values in everyday life. Scores can range from 1 to 100 with higher scores indicating greater contact with values in everyday life, which is generally considered desirable and a sign of good functioning.
Time Frame: Pre-treatment, and one- and three-month follow-ups
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment as Usual Plus ACT | Treatment as Usual
Number analyzed (Participants) | 34 | 33
score on a scale
  Pre-treatment | 34.3 [27.32 to 41.28] | 30.38 [22.59 to 38.17]
  One-Month Follow-up: number analyzed (Participants) | 20 | 23
  One-Month Follow-up | 46.10 [37.03 to 55.17] | 37.72 [28.91 to 46.54]
  Three-Month Follow-up: number analyzed (Participants) | 20 | 18
  Three-Month Follow-up | 41.94 [33.58 to 50.31] | 38.03 [27.22 to 48.84]

6. Secondary Outcome: Inventory of Psychosocial Functioning (Used to Assess Change)
Description: Self-report measure that assesses impairment within the last 30 days across a spectrum of psychosocial domains. Will be examined as a candidate outcome measure for a future efficacy trial. Response options range from 0 = never to 6 = always. The measure yields a mean score for the total scale. Higher scores indicate less functional impairment. The total scale score is reported.
Time Frame: Pre-treatment, and one- and three-month follow-ups
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment as Usual Plus ACT | Treatment as Usual
Number analyzed (Participants) | 35 | 35
units on a scale
  Pre-treatment | 2.89 [2.32 to 3.16] | 2.96 [2.66 to 3.26]
  One-month Follow-up: number analyzed (Participants) | 20 | 23
  One-month Follow-up | 2.02 [1.46 to 2.57] | 2.39 [2.07 to 2.71]
  Three-month Follow-up: number analyzed (Participants) | 20 | 19
  Three-month Follow-up | 2.01 [1.49 to 2.54] | 2.69 [2.35 to 3.03]

7. Secondary Outcome: PROMIS Global Short Form v1.1 (Used to Assess Change)
Description: Self-report measure assessing multiple domains of health. The scale yields two subscales: Global Physical Health and Global Mental Health. Global Mental Health will be examined as a candidate outcome measure for a future efficacy trial. The Global Mental Health sum score can range from 4 to 20, with higher scores indicating greater mental health.
Time Frame: Pre-treatment, and one- and three-month follow-ups
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment as Usual Plus ACT | Treatment as Usual
Number analyzed (Participants) | 34 | 34
score on a scale
  Pre-treatment | 9.41 [8.70 to 10.12] | 9.47 [8.78 to 10.16]
  One-month Follow-up: number analyzed (Participants) | 20 | 23
  One-month Follow-up | 11.20 [10.10 to 12.30] | 10.00 [9.00 to 11.00]
  Three-month Follow-up: number analyzed (Participants) | 20 | 19
  Three-month Follow-up | 10.75 [9.66 to 11.84] | 10.53 [9.52 to 11.53]

8. Secondary Outcome: PROMIS Short Form v2.0- Satisfaction With Social Roles and Activities 8a (Used to Assess Change)
Description: Self-report measure that assesses satisfaction with respondents' ability to perform various social activities. Will be examined as a candidate outcome measure for a future efficacy trial. Scale scores range from 8 to 40 with higher scores indicating greater satisfaction with ability to perform social activities.
Time Frame: Pre-treatment, and one- and three-month follow-ups
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment as Usual Plus ACT | Treatment as Usual
Number analyzed (Participants) | 34 | 33
units on a scale
  Pre-treatment | 18.15 [15.56 to 20.73] | 17.85 [15.58 to 20.11]
  One-month Follow-up: number analyzed (Participants) | 20 | 23
  One-month Follow-up | 22.90 [19.34 to 26.46] | 20.48 [17.60 to 23.36]
  Three-month Follow-up: number analyzed (Participants) | 20 | 19
  Three-month Follow-up | 23.10 [19.03 to 27.17] | 20.63 [17.31 to 23.94]

9. Secondary Outcome: Columbia Suicide-Severity Rating Scale (Used to Assess Change)
Description: Clinician-administered interview that assesses suicidal ideation and behavior. Will be examined as a candidate outcome measure for a future efficacy trial. Suicidal ideation intensity scores can range from 0 to 25 with higher scores indicating a greater intensity of suicidal ideation. Suicidal ideation intensity scale scores are reported.
Time Frame: Pre-treatment, and one- and three-month follow-ups
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment as Usual Plus ACT | Treatment as Usual
Number analyzed (Participants) | 35 | 35
units on a scale
  Pre-treatment | 15.37 [13.35 to 17.40] | 16.12 [14.06 to 18.18]
  One-month Follow-up: number analyzed (Participants) | 20 | 23
  One-month Follow-up | 6.75 [3.23 to 10.27] | 6.22 [2.96 to 9.47]
  Three-month Follow-up: number analyzed (Participants) | 23 | 19
  Three-month Follow-up | 3.52 [0.89 to 6.16] | 8.11 [4.18 to 12.03]

ADVERSE EVENTS:
Time Frame: One year, seven months
Arm/Group | Treatment as Usual Plus ACT | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

LIMITATIONS AND CAVEATS:
Outcome data are provided, but should not be used to draw conclusions about the efficacy of ACT for Life given recommendations for pilot study best practices (e.g., Eldrige et al., 2016) and data lost to follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/83/NCT02751983/Prot_SAP_000.pdf